CLINICAL TRIAL: NCT05297149
Title: Effect of Hippotherapy on Balance, Functional Mobility, and Functional Independence in Children With Down Syndrome: A Randomized Controlled Trial
Brief Title: Effect of Hippotherapy in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Seda Saka, PT PhD, Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ssaka4
Record Dates: First submitted 2022-03-04; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Down Syndrome
Keywords: Hippotherapy; Functional Mobility; Balance; Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hippotherapy group (Experimental): Participants that are performed hippotherapy
  Interventions: Behavioral: Hippotherapy
- Control group (Active Comparator): Participants that are performed home exercise program
  Interventions: Behavioral: Home exrecises

INTERVENTIONS:
Behavioral: Hippotherapy — The hippotherapy program consisted of 6 weekly sessions that varied in duration between 20 and 30 minutes depending on the weekly program and the participant's condition. Each session started with brief greetings and contact with the horse.
  Arms: hippotherapy group
Behavioral: Home exrecises — The home exercise program consisted of the following balance training exercises: one leg standing on foam with eyes open and closed, double leg standing on foam with eyes open and closed, walking in tandem with eyes open and closed, balance exercises on an inclined surface, balance exercises in squat, and jumping over an obstacle on the ground. All participants performed the exercises under parental supervision, 3 times per week for 6 weeks. The physiotherapist made video calls to the children and parents to ensure their adherence to the home exercise program.
  Arms: Control group

SUMMARY:
Purpose: The aim of this study was to determine the effect of hippotherapy on balance, functional mobility, and functional independence in children with Down syndrome (DS).

Methods: Thirty-four children with DS were randomly assigned to the experimental (hippotherapy) and control groups after initial assessment. Both groups received physiotherapy including balance exercises, and the experimental group also received hippotherapy. Pediatric Balance Scale (PBS), Timed Up and Go Test (TUG), and Functional Independence Measure for Children (WeeFIM) were used before and after the intervention.

DETAILED DESCRIPTION:
Purpose: The aim of this study was to determine the effect of hippotherapy on balance, functional mobility, and functional independence in children with Down syndrome (DS).

Methods: Thirty-four children with DS were randomly assigned to the experimental (hippotherapy) and control groups after initial assessment. Both groups received physiotherapy including balance exercises, and the experimental group also received hippotherapy. Pediatric Balance Scale (PBS), Timed Up and Go Test (TUG), and Functional Independence Measure for Children (WeeFIM) were used before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with down syndrome
* being aged 4 to 14 years
* being voluntary

Exclusion Criteria:

* having a history of previous hippotherapy intervention,
* having a phobia related to horse riding, epileptic seizures, atlantoaxial instability, and
* having any orthopedic, neurological, or cardiovascular disease that prevents physical activity.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale (PBS) | Change from baseline PBS at 6th week
  The PBS is a modified version of the Berg Balance Scale that is used to assess functional balance skills in children with mild to moderate motor impairment. The scale consists of 14 items that are scored from 0 (lowest function) to 4 (highest function) with a maximum score of 56 points. Lower scores indicate poorer balance. The PBS has been validated for use in children with neuromotor dysfunction.
Timed Up and Go Test (TUG) | Change from baseline TUG at 6th week
  The TUG assesses balance and functional mobility. The time required for the person to stand up from a chair, walk 3 meters forward, return to the chair, and sit down again was recorded. Times of 14 seconds or more are interpreted as high risk of falling. The TUG was reported to be reliable for assessing functional mobility in people with DS.
Pediatric Functional Independence Measure for Children (WeeFIM) | Change from baseline WeeFIM at 6th week
  The WeeFIM is a pediatric version of the Functional Independence Measure (FIM) that was developed to measures a child's consistent functional performance in essential daily functional skills (independence in self-care, sphincter control, transfers, locomotion, communication, and social cognition). It is an 18-item, 7-level ordinal scale instrument (score range: 18-126) and can be used for children with developmental disabilities aged 6 months to 21 years.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, PT, PhD, Study Director — Haliç University
Locations (1):
- Haliç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bronson C, Brewerton K, Ong J, Palanca C, Sullivan SJ. Does hippotherapy improve balance in persons with multiple sclerosis: a systematic review. Eur J Phys Rehabil Med. 2010 Sep;46(3):347-53. Epub 2010 Apr 13. PMID 20927000
- [Result] Moriello G, Terpstra ME, Earl J. Outcomes following physical therapy incorporating hippotherapy on neuromotor function and bladder control in children with Down syndrome: A case series. Phys Occup Ther Pediatr. 2020;40(3):247-260. doi: 10.1080/01942638.2019.1615601. Epub 2019 May 20. PMID 31106675
- [Result] Portaro S, Cacciola A, Naro A, Cavallaro F, Gemelli G, Aliberti B, De Luca R, Calabro RS, Milardi D. Can Individuals with Down Syndrome Benefit from Hippotherapy? An Exploratory Study on Gait and Balance. Dev Neurorehabil. 2020 Aug;23(6):337-342. doi: 10.1080/17518423.2019.1646830. Epub 2019 Jul 25. PMID 31342817